CLINICAL TRIAL: NCT00928070
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Trial To Evaluate The Efficacy And Safety Of Fesoterodine Flexible Dose Regimen In Vulnerable Elderly Patients With Overactive Bladder.
Brief Title: A Study Of Efficacy And Safety Of Fesoterodine In Vulnerable Elderly Subjects With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0221049
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2012-12

CONDITIONS: Overactive Bladder
Keywords: Urgency Urinary Incontinence OAB
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fesoterodine (Experimental)
  Interventions: Drug: Fesoterodine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine 4 mg and 8 mg
  Arms: Fesoterodine
Drug: Placebo — Placebo sham 4 mg and 8 mg
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy and safety of a flexible dose regimen of fesoterodine on urgency urinary incontinence (UUI) episodes in vulnerable elderly subjects with overactive bladder (OAB).

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects 65 years of age or older
* OAB symptoms for at least 3 months
* score 3 or greater on Vulnerable Elderly Survey (VES-13)
* adequate mobility for independent toileting
* mean number of at least 2 UUI episodes per 24 hours
* mean urinary frequency of 8 or more micturitions per 24 hours
* able to independently complete the bladder diaries

Exclusion Criteria:

* PVR urinary volume greater than 200 ml
* MMSE score less than 20
* greater than 15 UUI episodes per 24 hours
* creatinine clearance less than 30 ml/min
* an average resting heart rate of greater than or equal to 90 beats per minute

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 566 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (109):
- United States (109):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Green Valley, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Tuscon, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Fairfield, California
  - Pfizer Investigational Site, Glendora, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Mission Viejo, California
  - Pfizer Investigational Site, Murrieta, California
  - Pfizer Investigational Site, Norwalk, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Rancho Santa Margarita, California
  - Pfizer Investigational Site, San Bernardino, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Vacaville, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Parker, Colorado
  - Pfizer Investigational Site, Groton, Connecticut
  - Pfizer Investigational Site, Milford, Connecticut
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Bonita Springs, Florida
  - Pfizer Investigational Site, Boynton Beach, Florida
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Plant City, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Trinity, Florida
  - Pfizer Investigational Site, Wellington, Florida
  - Pfizer Investigational Site, Winter Haven, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Arkansas City, Kansas
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Glen Burnie, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Picayune, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Moorestown, New Jersey
  - Pfizer Investigational Site, Sewell, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Willoughby Hills, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Erie, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Leander, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Burien, Washington
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Dubeau CE, Kraus SR, Griebling TL, Newman DK, Wyman JF, Johnson TM 2nd, Ouslander JG, Sun F, Gong J, Bavendam T. Effect of fesoterodine in vulnerable elderly subjects with urgency incontinence: a double-blind, placebo controlled trial. J Urol. 2014 Feb;191(2):395-404. doi: 10.1016/j.juro.2013.08.027. Epub 2013 Aug 21. PMID 23973522
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221049&StudyName=A%20Study%20Of%20Efficacy%20And%20Safety%20Of%20Fesoterodine%20In%20Vulnerable%20Elderly%20Subjects%20With%20Overactive%20Bladder

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to fesoterodine 4 milligram (mg) oral tablet once daily for 4 weeks followed by placebo matched to fesoterodine 8 mg once daily as part of optional dose escalation at investigator's discretion for remaining 8 weeks.
- Fesoterodine: Fesoterodine 4 mg oral tablet once daily for 4 weeks followed by an optional dose-escalation to 8 mg once daily at investigator's discretion for remaining 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Fesoterodine
Started | 283 | 283
Treated | 281 | 281
Completed | 220 | 226
Not Completed | 63 | 57
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Adverse Event | 14 | 26
Not completed — Lack of Efficacy | 9 | 5
Not completed — Did not meet entrance criteria | 16 | 9
Not completed — Protocol Violation | 6 | 5
Not completed — Randomized but not treated | 2 | 2
Not completed — Other | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants who received placebo matched to fesoterodine 4 milligram (mg) oral tablet once daily for 4 weeks followed by placebo matched to fesoterodine 8 mg once daily as part of optional dose escalation at investigator's discretion for remaining 8 weeks.
- Fesoterodine: Participants who received fesoterodine 4 mg oral tablet once daily for 4 weeks followed by an optional dose-escalation to 8 mg once daily at investigator's discretion for remaining 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fesoterodine | Total
Number analyzed (Participants) | 281 | 281 | 562
Age, Customized [Number; unit: participants]
  65 to 74 years | 134 | 145 | 279
  75 to 84 years | 118 | 106 | 224
  At least 85 years | 29 | 30 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 225 | 461
  Male | 45 | 56 | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours
Description: UUI episodes were defined as those with the Urinary Sensation Scale (USS) rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline
Population: Full analysis set (FAS) population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. 'N' (number of participants analyzed) signifies those participants who had baseline UUI episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 250 | 256
episodes per 24 hours | 3.93 (2.16) | 4.07 (2.33)

2. Primary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 12
Description: UUI episodes were defined as those with the USS rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Week 12
Population: FAS population. Last observation carried forward (LOCF) method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline UUI episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 250 | 256
episodes per 24 hours | -2.20 (0.15) | -2.84 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Analysis of covariance (ANCOVA) model with terms for treatment, center, centered baseline, and centered baseline by treatment interaction was used to calculate p-value; Test type: Superiority or Other; p = 0.0018, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -0.65, 95% CI 2-sided [-1.05 to -0.24], Standard Error of Mean 0.21

3. Secondary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 4
Description: as for outcome 2
Time Frame: Baseline, Week 4
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline UUI episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 4.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 248 | 255
episodes per 24 hours | -1.54 (0.16) | -2.36 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; ANCOVA model with terms for treatment, center, centered baseline, and centered baseline by treatment interaction was used to calculate p-value; Test type: Superiority or Other; p = 0.0003, ANCOVA — Statistical testing, two-sided, was done at 5% significance level; Least squares mean difference = -0.82, 95% CI 2-sided [-1.27 to -0.38], Standard Error of Mean 0.23

4. Secondary Outcome: Percent Change From Baseline in Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 4 and 12
Description: Percent change of UUI episodes per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (i.e., 100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline UUI episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 250 | 256
percent change
  Change at Week 4 | -39.2 (65.7) | -57.2 (54.4)
  Change at Week 12 | -55.4 (63.1) | -71.2 (51.4)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: Ranked ANCOVA model with terms for treatment and center with ranked baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, Ranked ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Testing for percent change from baseline was only carried out for given endpoint if corresponding numeric change result was statistically significant
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 12: Ranked ANCOVA model with terms for treatment and center with ranked baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0001, Ranked ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Mean Number of Micturitions Per 24 Hours
Description: Micturitions include episodes of voluntary micturition and episodes of UUI. UUI episodes were defined as those micturitions with USS rating of 5 in the diary in participants with UUI at baseline. USS rating 5: Unable to hold; leak urine.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline micturition frequency greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 253 | 258
micturitions per 24 hours | 12.22 (3.21) | 12.11 (3.06)

6. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 4 and 12
Description: as for outcome 5
Time Frame: Baseline, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline micturition frequency greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: micturitions per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 253 | 258
micturitions per 24 hours
  Change at Week 4 | -0.77 (0.17) | -1.64 (0.17)
  Change at Week 12 | -1.50 (0.16) | -2.34 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: ANCOVA model with terms for treatment and center with centered baseline as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0003, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -0.87, 95% CI 2-sided [-1.35 to -0.40], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 12: ANCOVA model with terms for treatment and center with centered baseline as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0003, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -0.84, 95% CI 2-sided [-1.29 to -0.39], Standard Error of Mean 0.23

7. Secondary Outcome: Percent Change From Baseline in Micturitions Per 24 Hours at Week 4 and 12
Description: Percent change of micturitions per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (i.e., 100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4, 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 253 | 258
percent change
  Change at Week 4 | -5.1 (24.4) | -12.7 (19.1)
  Change at Week 12 | -10.4 (22.4) | -17.8 (19.6)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Ranked ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.0001, Ranked ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; [statistical method as in outcome 4, analysis 1]

8. Secondary Outcome: Mean Number of Micturition-related Urgency Episodes Per 24 Hours
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of greater than or equal to (>=) 3 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 256
episodes per 24 hours | 10.30 (3.67) | 10.02 (3.54)

9. Secondary Outcome: Change From Baseline in Mean Number of Micturition-related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: as for outcome 8
Time Frame: Baseline, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 256
episodes per 24 hours
  Change at Week 4 | -1.64 (0.24) | -2.74 (0.24)
  Change at Week 12 | -2.75 (0.25) | -4.15 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0014, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -1.10, 95% CI 2-sided [-1.77 to -0.43], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 12: ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -1.40, 95% CI 2-sided [-2.10 to -0.70], Standard Error of Mean 0.35

10. Secondary Outcome: Percent Change From Baseline in Micturition-related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Percent change of micturition-related urgency episodes per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (i.e., 100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4, 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 256
percent change
  Change at Week 4 | -12.7 (45.0) | -26.2 (39.4)
  Change at Week 12 | -23.9 (46.4) | -39.7 (45.0)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, Ranked ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.0001, Ranked ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; [statistical method as in outcome 4, analysis 1]

11. Secondary Outcome: Mean Number of Nocturnal Micturition-related Urgency Episodes Per 24 Hours
Description: Nocturnal micturition-related urgency episodes had USS rating of 3 or more that occurred between time participant went to bed and time he or she arose to start next day. Number of nocturnal micturition-related urgency episodes per 24 hours was calculated as sum of all nocturnal micturition-related urgency episodes divided by total number of diary days collected at that visit.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 254
episodes per 24 hours | 2.87 (1.51) | 2.69 (1.38)

12. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Micturition-related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: as for outcome 11
Time Frame: Baseline, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline nocturnal urgency episodes greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 254
episodes per 24 hours
  Change at Week 4 | -0.44 (0.09) | -0.58 (0.09)
  Change at Week 12 | -0.68 (0.09) | -0.97 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.2511, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -0.15, 95% CI 2-sided [-0.39 to 0.10], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.0189, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -0.29, 95% CI 2-sided [-0.53 to -0.05], Standard Error of Mean 0.12

13. Secondary Outcome: Percent Change From Baseline in Nocturnal Micturition-related Urgency Episodes Per 24 Hours at Week 4 and 12
Description: Percent change of nocturnal micturition-related urgency episodes per 24 hours was calculated as change in 24-hour mean at that visit divided by the baseline 24-hour mean multiplied by 100 (i.e., 100*(Week 4 or 12 - baseline)/baseline).
Time Frame: Baseline, Week 4, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 254
percent change
  Change at Week 4 | -4.9 (68.2) | -18.0 (62.6)
  Change at Week 12 | -15.5 (63.6) | -31.2 (59.5)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.0010, Ranked ANCOVA — Statistical testing, two-sided, was done at 5% significance level; [statistical method as in outcome 4, analysis 1]

14. Secondary Outcome: Frequency-Urgency Sum Rating Per 24 Hours
Description: Frequency-urgency sum is total USS ratings recorded for all micturitions in 24-hour day. Number of USS ratings per 24 hours is sum of all USS ratings divided by the total diary days collected at that visit. USS scale: 1=No feeling of urgency to 5=Unable to hold: leak urine.
Time Frame: Baseline
Population: FAS population. Here, 'N' (number of participants analyzed) signifies those participants who had baseline frequency urgency sum rating greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 256
units on a scale | 45.33 (13.20) | 44.92 (13.45)

15. Secondary Outcome: Change From Baseline in Frequency-Urgency Sum Rating Per 24 Hours at Week 4 and 12
Description: Frequency-urgency sum is total USS ratings recorded for all micturitions in 24-hour day. Number of USS ratings per 24 hours is sum of all USS ratings divided by the total diary days collected at that visit. USS scale: 1=No feeling of urgency to 5=Unable to hold: leak urine. Numerical decrease indicates improvement.
Time Frame: Baseline, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had baseline frequency urgency sum rating greater than 0 per 24 hours and non-missing change from baseline value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 251 | 256
units on a scale
  Change at Week 4 | -6.95 (0.86) | -11.62 (0.86)
  Change at Week 12 | -11.53 (0.84) | -16.50 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -4.67, 95% CI 2-sided [-7.04 to -2.30], Standard Error of Mean 1.21
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -4.97, 95% CI 2-sided [-7.27 to -2.66], Standard Error of Mean 1.17

16. Secondary Outcome: Change From Baseline in Mean Number of Protective Undergarments Changed Due to Urinary Leakage Per 24 Hours at Week 4 and 12
Description: Protective Undergarments included pads, protective padding, protective underwear (pull up), and briefs (diaper). The mean number of undergarments changed per 24 hours was calculated as the total number of undergarments changed divided by the total number of diary days collected at that visit. Change from baseline values were reported at week 4 for subsets of population with baseline values less than or equal to (=<) 3.5 and more than (>) 3.5 undergarments/day and at Week 12 for subsets of population with baseline values =< 2.5 and > 2.5 undergarments/day.
Time Frame: Baseline, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'n' is signifying those participants of the population subsets who were evaluated for this measure at the time point for each group respectively.
Measure: Mean (Standard Deviation); unit: undergarments
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 281 | 281
undergarments
  Baseline: =<3.5 undergarments (n=193,184) | 1.41 (0.84) | 1.49 (0.74)
  Baseline: >3.5 undergarments (n=12,19) | 4.97 (1.84) | 4.81 (0.92)
  Baseline: =<2.5 undergarments (n=172,169) | 1.21 (0.63) | 1.35 (0.62)
  Baseline: >2.5 undergarments (n=35,35) | 3.71 (1.42) | 3.94 (1.18)
  Change at Week 4: =<3.5 undergarments(n=193,184) | -0.27 (1.13) | -0.61 (1.09)
  Change at Week 4: >3.5 undergarments(n=12,19) | -2.56 (3.07) | -2.11 (3.38)
  Change at Week 12: =<2.5 undergarments(n=172,169) | -0.31 (1.06) | -0.72 (0.82)
  Change at Week 12: >2.5 undergarments(n=35,35) | -2.14 (2.06) | -1.98 (1.86)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: =<3.5 undergarments- Protective undergarment usage was analyzed to compare treatments on separate subsets, based on baseline protective undergarment use (=<3.5/day and >3.5/day), using a 2 sample t-test. This method was applied because there was a statistically significant qualitative baseline by treatment interaction; Test type: Superiority or Other; p = 0.0035, t-test, 2 sided — Statistical testing, two-sided, was done at 5% alpha level; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.56 to -0.11], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 4: >3.5 undergarments- Protective undergarment usage was analyzed to compare treatments on separate subsets, based on baseline protective undergarment use (=<3.5/day and >3.5/day), using a 2 sample t-test. This method was applied because there was a statistically significant qualitative baseline by treatment interaction; Test type: Superiority or Other; p = 0.7089, t-test, 2 sided — Statistical testing, two-sided, was done at 5% alpha level; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-2.01 to 2.92], Standard Error of Mean 1.21
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Change at Week 12: =<2.5 undergarments- Protective undergarment usage was analyzed to compare treatments on separate subsets, based on baseline protective undergarment use (=<2.5/day and >2.5/day), using a 2 sample t-test. This method was applied because there was a statistically significant qualitative baseline by treatment interaction; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Statistical testing, two-sided, was done at 5% alpha level; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.61 to -0.21], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Change at Week 12: >2.5 undergarments- Protective undergarment usage was analyzed to compare treatments on separate subsets, based on baseline protective undergarment use (=<2.5/day and >2.5/day), using a 2 sample t-test. This method was applied because there was a statistically significant qualitative baseline by treatment interaction; Test type: Superiority or Other; p = 0.7437, t-test, 2 sided — Statistical testing, two-sided, was done at 5% alpha level; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.78 to 1.09], Standard Error of Mean 0.47

17. Secondary Outcome: Percentage of Participants With Change From Screening in Patient Perception of Bladder Condition (PPBC) at Week 4 and 12
Description: PPBC: a self-administered, single-item, questionnaire that asks participants to describe their perception of their bladder-related problems. The PPBC assessment is rated on a 6-point scale: 1=no problems at all, 2=some very minor problems, 3=some minor problems, 4=moderate problems, 5=severe problems, 6=many severe problems. Deterioration=score difference is greater than 0; no change=score difference is 0; minor improvement=score difference is -1; major difference=score difference is less than or equal to -2.
Time Frame: Screening, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing change from baseline value at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 264 | 265
percentage of participants
  Baseline: No problems at all | 0.0 | 0.0
  Baseline: Some very minor problems | 0.0 | 0.0
  Baseline: Some minor problems | 0.0 | 0.0
  Baseline: Moderate problems | 44.7 | 44.5
  Baseline: Severe problems | 43.9 | 44.2
  Baseline: Many severe problems | 11.4 | 11.3
  Change at Week 4: Deterioration | 12.3 | 9.5
  Change at Week 4: No change | 42.5 | 29.8
  Change at Week 4: Minor improvement | 25.3 | 27.5
  Change at Week 4: Major improvement | 19.9 | 33.2
  Change at Week 12: Deterioration | 12.1 | 7.2
  Change at Week 12: No change | 33.7 | 27.2
  Change at Week 12: Minor improvement | 25.0 | 26.8
  Change at Week 12: Major improvement | 29.2 | 38.9
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4- deterioration, no change, minor improvement and major improvement: Cochran-Mantel-Haenszel (CMH) test with modified ridit scoring controlling for center was used to calculate p-value; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — Statistical testing, two-sided, was done at 5% alpha level
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 12- deterioration, no change, minor improvement and major improvement: CMH test with modified ridit scoring controlling for center was used to calculate p-value; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel — Statistical testing, two-sided, was done at 5% alpha level

18. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score
Description: OAB-q: a self-administered, 33-item, questionnaire that assesses how much the participant has been bothered by selected bladder symptoms. Each item rated by participant on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Symptom bother score derived as sum of scores for questions 1-8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/range]*100. Higher scores values indicative of greater symptom bother.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing change from baseline value at both Weeks 4 and 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 267 | 269
units on a scale | 67.67 (18.59) | 67.25 (19.04)

19. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score at Week 4 and 12
Description: as for outcome 18
Time Frame: Baseline, Week 4, 12
Population: FAS population. LOCF method was used to impute only Week 12 missing data but not Week 4 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing change from baseline value at both Weeks 4 and 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 267 | 269
units on a scale
  Change at Week 4 | -13.81 (1.46) | -22.96 (1.46)
  Change at Week 12 | -20.48 (1.58) | -28.08 (1.58)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -9.15, 95% CI 2-sided [-12.85 to -5.45], Standard Error of Mean 1.88
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -7.60, 95% CI 2-sided [-11.60 to -3.61], Standard Error of Mean 2.03

20. Secondary Outcome: Health Related Quality of Life (HRQL) Domain and Total Score of Overactive Bladder Questionnaire (OAB-q)
Description: OAB-q: self-administered, 33-item, questionnaire, assesses how much participant has been bothered by selected bladder symptoms. Each item rated on Likert scale 1 (least symptom bother) to 6 (most symptom bother). Questions 9 to 33 constitute HRQL, includes domains: concern, coping, sleep, and social function. HRQL domain and total raw score derived as sum of scores. Transformed score range 0 to 100 (Total HRQL or domain) = [(Highest possible raw score-Actual total raw score)/Raw score range]*100. Higher transformed scores indicative of better HRQL.
Time Frame: Baseline
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing change from baseline value at both Week 4 and 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 267 | 269
units on a scale
  Concern domain | 45.89 (25.38) | 46.57 (25.88)
  Coping domain | 44.72 (26.12) | 44.74 (26.76)
  Sleep domain | 40.19 (26.51) | 43.41 (25.76)
  Social interaction domain | 72.05 (25.35) | 72.70 (25.45)
  Total | 49.61 (22.35) | 50.58 (22.87)

21. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL) Domain and Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 4 and 12
Description: as for outcome 20
Time Frame: Baseline, Week 4, 12
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. LOCF method was used to impute Week 12 missing data. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing change from baseline value at both Week 4 and 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 267 | 269
units on a scale
  Change at Week 4: concern domain | 12.35 (1.61) | 20.51 (1.61)
  Change at Week 4: coping domain | 12.90 (1.65) | 19.86 (1.66)
  Change at Week 4: sleeping domain | 13.33 (1.56) | 17.33 (1.56)
  Change at Week 4: social interaction domain | 8.77 (1.19) | 11.22 (1.19)
  Change at Week 4: total | 12.00 (1.37) | 17.80 (1.38)
  Change at Week 12: concern domain | 17.20 (1.70) | 26.24 (1.70)
  Change at Week 12: coping domain | 20.34 (1.72) | 25.66 (1.72)
  Change at Week 12: sleeping domain | 19.05 (1.63) | 23.10 (1.63)
  Change at Week 12: social interaction domain | 12.12 (1.26) | 14.47 (1.26)
  Change at Week 12: total | 17.55 (1.46) | 23.08 (1.46)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: concern domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 8.17, 95% CI 2-sided [4.09 to 12.25], Standard Error of Mean 2.08
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 4: coping domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0012, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 6.96, 95% CI 2-sided [2.77 to 11.15], Standard Error of Mean 2.13
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Change at Week 4: sleep domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0472, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 4.00, 95% CI 2-sided [0.05 to 7.95], Standard Error of Mean 2.01
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Change at Week 4: social interaction domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.1087, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 2.46, 95% CI 2-sided [-0.55 to 5.46], Standard Error of Mean 1.53
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Change at Week 4: total- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0012, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 5.79, 95% CI 2-sided [2.31 to 9.28], Standard Error of Mean 1.77
Statistical Analysis 6: Comparison: Placebo vs Fesoterodine; Change at Week 12: concern domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 9.04, 95% CI 2-sided [4.75 to 13.33], Standard Error of Mean 2.19
Statistical Analysis 7: Comparison: Placebo vs Fesoterodine; Change at Week 12: coping domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0169, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 5.32, 95% CI 2-sided [0.96 to 9.67], Standard Error of Mean 2.22
Statistical Analysis 8: Comparison: Placebo vs Fesoterodine; Change at Week 12: sleep domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0546, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 4.05, 95% CI 2-sided [-0.08 to 8.17], Standard Error of Mean 2.10
Statistical Analysis 9: Comparison: Placebo vs Fesoterodine; Change at Week 12: social interaction domain- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.1497, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 2.35, 95% CI 2-sided [-0.85 to 5.55], Standard Error of Mean 1.63
Statistical Analysis 10: Comparison: Placebo vs Fesoterodine; Change at Week 12: total- ANCOVA model with terms for treatment and center with centered baseline value as a covariate was used to calculate p-value; Test type: Superiority or Other; p = 0.0034, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = 5.53, 95% CI 2-sided [1.84 to 9.23], Standard Error of Mean 1.88

22. Secondary Outcome: Overactive Bladder Satisfaction Questionnaire (OAB-S) Total Score on Satisfaction With OAB Control
Description: OAB-S: a validated self-administered instrument that evaluates OAB medication expectations, daily life with AB, and satisfaction with OAB medication and includes 3 stand-alone items that assess overall expectation, satisfaction, and willingness to continue treatment. Satisfaction coded on scale of 1 to 5: (1=very satisfied to 5=very dissatisfied). Coding reversed algorithmically and results transformed: total score range 0 to100. Higher final response value associated with better satisfaction.
Time Frame: Week 12
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing value at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 224 | 228
units on a scale | 52.98 (33.82) | 68.89 (28.89)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; ANOVA model with treatment and center as factors was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, ANOVA — Statistical testing, two-sided, was done at 5% significance level; Least squares mean difference = 16.25, 95% CI 2-sided [10.43 to 22.08], Standard Error of Mean 2.96

23. Secondary Outcome: Percentage of Participants With Overactive Bladder Satisfaction Questionnaire (OAB-S) Global Medication Satisfaction Question Response
Description: Participant's response to question, "overall, how satisfied are you with your OAB medication?" was obtained on a 5 point scale, 1- very satisfied, 2- somewhat satisfied, 3- neither dissatisfied nor satisfied, 4- somewhat dissatisfied and 5- very dissatisfied. Response values 1 and 2 were combined into "satisfied", and 4 and 5 were combined into "dissatisfied".
Time Frame: Week 12
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 224 | 227
percentage of participants
  Not satisfied | 37.5 | 18.9
  Neither dissatisfied nor satisfied | 15.2 | 9.3
  Satisfied | 47.3 | 71.8
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Not satisfied, neither dissatisfied nor satisfied, satisfied: CMH test with modified ridit scoring controlling for center was used; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Statistical testing, two-sided, was done at 5% alpha level

24. Secondary Outcome: Mini Mental State Examination (MMSE)
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranges from 0 to 30, higher score indicates better cognitive state.
Time Frame: Screening
Population: FAS population included all participants who received at least 1 dose of study drug and had at least 1 baseline or post-baseline efficacy assessment. Here, 'N' (number of participants analyzed) signifies those participants who had non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 220 | 223
units on a scale | 28.04 (2.05) | 28.16 (1.80)

25. Secondary Outcome: Change From Screening in Mini Mental State Examination (MMSE) Score at Week 12
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranges from 0 to 30, higher score indicates better cognitive state. Change: mean score at Week X minus mean score at baseline
Time Frame: Screening, Week 12
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 220 | 223
units on a scale | 0.33 (0.12) | 0.15 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; ANCOVA model with terms for treatment, center, centered baseline value, and centered baseline by treatment interaction; Test type: Superiority or Other; p = 0.2788, ANCOVA — Statistical testing, two-sided, was done at 5% alpha level; Least squares mean difference = -0.18, 95% CI 2-sided [-0.51 to 0.15], Standard Error of Mean 0.17

26. Secondary Outcome: Change From Baseline in Post Void Residual (PVR) Volume at Week 4 and 12
Description: PVR volume is defined as volume of urine remaining in the bladder immediately after urination.
Time Frame: Baseline, Week 4, 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 266 | 271
mL
  Baseline | 26.51 (35.36) | 25.69 (34.28)
  Change at Week 4 | 1.83 (41.30) | 13.43 (57.70)
  Change at Week 12 | -2.98 (35.95) | 13.58 (60.22)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Change at Week 4: Van Elteren's test adjusted by baseline PVR quartile was used to calculate p-value. The median difference was based on Hodges-Lehmann estimate; Test type: Superiority or Other; p = 0.0021, Van Elteren's test — Statistical testing, two-sided, was done at 5% alpha level; Median Difference (Final Values) = 4.00, 95% CI 2-sided [0.00 to 8.00]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Change at Week 12: Van Elteren's test adjusted by baseline PVR quartile was used to calculate p-value. The median difference was based on Hodges-Lehmann estimate; Test type: Superiority or Other; p < 0.0001, Van Elteren's test — Statistical testing, two-sided, was done at 5% alpha level; Median Difference (Final Values) = 7.00, 95% CI 2-sided [3.00 to 11.00]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 6/281 | 8/281
Other Adverse Events (participants affected / at risk) | 120/281 | 155/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=281) | Fesoterodine (N=281)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=281) | Fesoterodine (N=281)
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Left atrial dilatation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Asthenopia (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 3 | 4
Eye discharge (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Eye oedema (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 5 | 0
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 12 | 31
Diarrhoea (Gastrointestinal disorders) | 7 | 8
Diverticulum (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 17 | 66
Dyspepsia (Gastrointestinal disorders) | 1 | 7
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Tongue dry (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 3 | 8
Gait disturbance (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 6 | 6
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Therapeutic response unexpected (General disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Allergy to chemicals (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 5 | 1
Candidiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 5 | 5
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 5
Staphylococcal infection (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 3
Urinary tract infection (Infections and infestations) | 10 | 6
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 7
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 2
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 2
Blood uric acid increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Nitrite urine present (Investigations) | 1 | 0
Residual urine volume increased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 5 | 7
Hypersomnia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 3
Sleep disorder (Psychiatric disorders) | 0 | 1
Bladder mass (Renal and urinary disorders) | 1 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 3 | 4
Haematuria (Renal and urinary disorders) | 1 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 9
Urine flow decreased (Renal and urinary disorders) | 1 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.